CLINICAL TRIAL: NCT00041600
Title: Human Epilepsy Genetics--Neuronal Migration Disorders Study
Status: Recruiting | Type: Observational
Sponsor: Harvard University Faculty of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Howard Hughes Medical Institute (Other)
Responsible Party: Principal Investigator, Dr. Chris Walsh, Investigator, Harvard University Faculty of Medicine
Other Study IDs: R01NS035129 (NIH)
Record Dates: First submitted 2002-07-11; First posted 2002-07-12 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Brain Malformation; Neuronal Migration Disorder; Cognition Disorder; Epilepsy
Keywords: epilepsy; seizures; disorders of human cognition; neuronal migration; neuronal migration disorders; lissencephaly; schizencephaly; polymicrogyria; heterotopia; microcephaly; pachygyria
MeSH Terms: conditions — Malformations of Cortical Development, Group II; Cognition Disorders; Epilepsy; Seizures; Lissencephaly; Schizencephaly; Polymicrogyria; Choristoma; Microcephaly

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — whole blood, DNA
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify genes responsible for epilepsy, brain malformations and disorders of human cognition.

DETAILED DESCRIPTION:
Epilepsy is responsible for tremendous long-term healthcare costs. Analysis of inherited epilepsy conditions has allowed for identification of several key genes active in the developing brain. Although many genetic abnormalities of the brain are rare and lethal, rapidly advancing knowledge of the structure of the human genome makes it a realistic goal to identify genes responsible for other epileptic conditions, related brain malformations and disorders of cognition.

The purpose of this study is to identify genes responsible for epilepsy and disorders of human cognition (EDHC). The Walsh Laboratory at Boston Children's Hospital is looking for genes involved in brain development. Conditions that we study include brain malformations, such as polymicrogyria, lissencephaly, pachygyria, heterotopias, microcephaly and cerebellar hypoplasia, and inherited disorders of cognition, such as familial intellectual disability and familial autism. People with these conditions also often have epilepsy. The structural brain abnormalities are usually diagnosed by brain MRI or sometimes CT scans. Adults and children with these conditions, and their family members, are invited to participate in our study. By comparing the DNA of individuals or families that carry EDHC to the DNA of people in the general population, it may be possible to learn more about the genetic bases of certain forms of EDHC.

Study participants must have a brain malformation or disorder of cognition, such as familial intellectual disability or autism, in order to take part in this research.

ELIGIBILITY:
INCLUSION:

* Males and females of any age.
* Persons with a brain malformation or disorder of cognition (familial intellectual disability [previously known as mental retardation] or autism).

EXCLUSION:

* Persons without a brain malformation or disorder of cognition (familial intellectual disability (previously known as mental retardation] or autism).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants will be selected through collaborations with clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 1996-04; Primary Completion 2030-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Identification and characterization of genes important in normal brain development and associated with brain malformations. | Ongoing
  Genetic variants associated with disorder of brain development

CONTACTS AND LOCATIONS:
Overall Officials: Christopher A. Walsh, M.D., Ph.D., Principal Investigator — Harvard Institutes of Medicine
Locations (1):
- Boston Children's Hospital, Walsh Laboratory, Boston, Massachusetts, United States

REFERENCES:
- See also: laboratory website — http://www.walshlab.org